CLINICAL TRIAL: NCT04536038
Title: The Effect of opt-in Versus Opt-out Framing on Clinical Trial Enrollment Among Patients With Peripheral Artery Disease
Brief Title: Framing Clinical Trial Enrollment for Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 842681
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opt-in (No Intervention): Patients randomized to opt-in framing will be instructed to visit the Way to Health website to enroll in the study, or to call or email the study coordinator with questions or for assistance in enrolling.
- Opt-out (Experimental): Patients randomized to opt-out framing will receive an email that frames participation in the study as part of the standard of care, and will be informed that a study coordinator will be calling them in the coming days to start enrollment in the study unless they opt out of participation.
  Interventions: Behavioral: Opt-out

INTERVENTIONS:
Behavioral: Opt-out — A study coordinator will call the patient unless they opt-out. See arm description for more details.
  Arms: Opt-out

SUMMARY:
It is uncertain whether opt-out framing will increase participation in a clinical trial intended to promote physical activity in patients with peripheral artery disease (PAD). This study will test whether opt-in or opt-out framing of study participation upon initial contact affects the proportion of patients who ultimately enroll in the study and the demographic characteristics of enrolled patients.

DETAILED DESCRIPTION:
The GAMEPAD study is a two-arm randomized controlled trial aimed at evaluating whether a home-based walking program with automated coaching augmented with gamification and behavioral economic principles improves functional capacity in patients with PAD. GAMEPAD will be conducted using the Way to Health platform, and patients will enroll and consent for participation online, with available help from a study coordinator by telephone. The present study will leverage the GAMEPAD enrollment process to test whether opt-in or opt-out framing of study participation upon initial contact affects the proportion of patients who ultimately enroll in the GAMEPAD study and the demographic characteristics of enrolled patients.

Eligible patients will be contacted via email to determine their interest in participation in the GAMEPAD study. Patients will be randomized 3:1 to an email message framing trial participation in a standard opt-in manner versus an email message framing trial participation in an opt-out manner.

Patients randomized to opt-in framing will be instructed to visit the Way to Health website to enroll in the GAME PAD study, or to call or email the study coordinator with questions or for assistance in enrolling. Patients randomized to opt-out framing will be informed that a study coordinator will be calling them in the coming days to discuss enrollment in the study.

Baseline characteristics of patients randomized to each framing method will be abstracted from the electronic health record and Penn Data Store, and will include age, sex, race/ethnicity, and medical comorbidities. Whether contacted patients created an account on the Way to Health website and/or ultimately consented for enrollment in the study will be captured.

For all outcomes, we will compare patients initially presented with study participation via opt-in framing versus opt-out framing. The primary outcome will be the proportion of patients that enroll in the GAMEPAD study. We will also report the proportion of enrolled patients that failed to complete the GAMEPAD study among those patients that ultimately enrolled.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have been seen in the University of Pennsylvania Health System
* Have an ICD-10 code consistent with peripheral artery disease (I70.2x, I70.3x-I70.7x, I73.9) or peripheral artery disease on their problem list
* Have an email address on file with the University of Pennsylvania Health System

Exclusion Criteria:

* Previously indicated unwillingness to be contacted by email for participation in research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5176 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opt-in | Opt-out
Started | 3909 | 1267
Completed | 3909 | 1267
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opt-in | Opt-out | Total
Number analyzed (Participants) | 3909 | 1267 | 5176
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (12.3) | 69.7 (12) | 69.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1589 | 523 | 2112
  Male | 2320 | 744 | 3064
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2622 | 882 | 3504
  Black | 916 | 289 | 1205
  Asian | 62 | 15 | 77
  Hispanic | 94 | 22 | 116
  Other | 215 | 59 | 274
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (6.5) | 29 (6.5) | 29.1 (6.5)
History of myocardial infarction [Count of Participants; unit: Participants] | 751 | 204 | 955
History of congestive heart failure [Count of Participants; unit: Participants] | 1353 | 430 | 1783
History of stroke or cerebrovascular event [Count of Participants; unit: Participants] | 1421 | 496 | 1917
History of dementia [Count of Participants; unit: Participants] | 101 | 46 | 147
History of pulmonary disease [Count of Participants; unit: Participants] | 1408 | 425 | 1833
History of Diabetes without complications [Count of Participants; unit: Participants] | 1620 | 508 | 2128
History of Diabetes with complications [Count of Participants; unit: Participants] | 818 | 248 | 1066
History of renal disease [Count of Participants; unit: Participants] | 1139 | 367 | 1506

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in GAMEPAD Intervention Study
Description: The proportion of patients that enroll in the GAMEPAD intervention study
Time Frame: Enrollment (period of approximately 6 months)
Population: The number of participants reported in the Participant Flow are participants that were active in the GAMEPAD trial. Participants Analyzed above are all the participants randomized to either opt in or opt out recruitment style that was contacted to be a part of the GAMEPAD Study.
Measure: Count of Participants; unit: Participants
Arm/Group | Opt-in | Opt-out
Number analyzed (Participants) | 3909 | 1267
Participants | 39 | 45

2. Other Pre Specified Outcome: Participants That Fail to Complete Study
Description: The proportion of patients enrolled in GAMEPAD that failed to complete the study
Time Frame: through the end of the 24-week study period
Measure: Number; unit: proportion of participants
Arm/Group | Opt-in | Opt-out
Number analyzed (Participants) | 39 | 45
proportion of participants | .154 | .067

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events were collected via participant reports through study surveys at 16 weeks, and 24-weeks or participant reports to study staff through text, email or phone call.
Arm/Group | Opt-in | Opt-out
All-Cause Mortality (participants affected / at risk) | 0/3909 | 1/1267
Serious Adverse Events (participants affected / at risk) | 1/3909 | 4/1267
Other Adverse Events (participants affected / at risk) | 14/3909 | 11/1267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opt-in (N=3909) | Opt-out (N=1267)
Orthopedic (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Cardiovascular (Cardiac disorders) | 0 (0) | 2 (3)
Fitbit-related (Product Issues) | 0 (0) | 0 (0)
Other (General disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opt-in (N=3909) | Opt-out (N=1267)
Orthopedic (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (4)
Cardiovascular (Cardiac disorders) | 1 (1) | 2 (2)
Fitbit-related (Product Issues) | 1 (1) | 1 (1)
Other (General disorders) | 8 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04536038/Prot_SAP_000.pdf